CLINICAL TRIAL: NCT01703585
Title: A Feasibility Study of Genomic Profiling Methods and Timing of Sample Collection to Evaluate Clonal Evolution and Tumor Heterogeneity
Brief Title: Feasibility Study of Genomic Profiling Methods and Timing in Tumor Samples
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: Ontario Institute for Cancer Research (Other); Princess Margaret Hospital, Canada (Other)
Responsible Party: Sponsor
Other Study IDs: MATCH-001
Record Dates: First submitted 2012-10-05; First posted 2012-10-10 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Colorectal Cancer; Breast Cancer; Gynecological Cancer; Metastatic; Eligible for Phase I or Phase II Study; Melanoma Cancer
Keywords: genomic analysis; genome; tumor; tissue; archival; biopsy; core needle; fine needle; DNA; gene; expression; sequencing
MeSH Terms: conditions — Colorectal Neoplasms; Breast Neoplasms; Neoplasm Metastasis; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fresh tumor tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- metastatic breast cancer
- metastatic colorectal cancer
- metastatic gynecological cancer
- metastatic melanoma

SUMMARY:
This is a feasibility study to look for genetic alterations in tissue and blood samples that may be useful in determining what treatments may be useful in the patient's cancer care.

DETAILED DESCRIPTION:
As part of the study, patients will have archival tumor tissue collected, and have tumor biopsies and blood samples taken. The samples will be tested for genetic alterations, and the results will be discussed with the patient including potential treatments. If patients agree, after they have received treatment for their cancer and their disease progresses, a second biopsy procedure will be done.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Histological or cytological proof of either metastatic breast, colorectal, gynecological or melanoma malignancy.
* At least one biopsiable lesion deemed medically accessible and safe to biopsy.
* Candidate for one or more phase I or II clinical trials at the time of study enrollment or at a later time point.
* Fulfills local institution's laboratory parameters for tumor biopsy.
* Willingness and ability of patient to provide signed voluntary informed consent.

Exclusion Criteria:

* Any condition that could interfere with a patient's ability to provide informed consent such as dementia or severe cognitive impairment.
* Any contraindication to undergoing a biopsy procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: metastatic breast, colorectal, gynecological cancer or melanoma
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2012-10-04 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Patient recruitment for paired core and fine needle biopsy greater than or equal to 50% of those screened or approached. | 2 years

SECONDARY OUTCOMES:
The rate of acceptable tumor samples from fresh core needle biopsy samples/total number of fresh core needle biopsy samples greater than or equal to 90% | 2 years
The rate of acceptable tumor samples from fresh fine needle biopsy samples/total number of fresh fine needle biopsy samples greater than or equal to 50% | 2 years
Successful analysis of fresh core needle biopsy samples and fresh fine needle biopsy samples greater than or equal to 50% | 2 years
  Sequenom or MiSeq/TSCAP and MiSeq/NGS
Analysis of fresh core needle biopsy samples and fresh fine needle biopsy samples from time from patient recruitment to final results, less than a defined period of time, in greater than or equal to 90% | 2 years
  Sequenom or MiSeq/TSCAP analysis from fresh core needle biopsy samples less than 4 weeks; sequenom or MiSeq/TSCAP analysis from fresh fine needle biopsy samples less than 8 weeks; MiSeq/NGS analysis from fresh core needle biopsy samples less than 8 weeks; MiSeq/NGS analysis from fresh fine needle biopsy samples less than 8 weeks
Actionable genomic result analysis of fresh core needle biopsy samples and fresh fine needle biopsy samples greater than or equal to 30% | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Lillian Siu, MD, Principal Investigator — Princess Margaret Cancer Centre; Bedard Philippe, MD, Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada